CLINICAL TRIAL: NCT03189485
Title: Tau PET Imaging in the NACC Study Cohort: Modulators of MTL Subregion Structure and Function in Normal and Pathological Aging
Brief Title: Tau PET Imaging in the NACC Study Cohort
Acronym: TPI
Status: Active, not recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, David Wolk, Co Director of the Penn Memory Center, University of Pennsylvania
Other Study IDs: 825944; R01AG055005 (NIH)
Record Dates: First submitted 2017-05-08; First posted 2017-06-16 (Actual); Last update posted 2025-10-29 (Actual); Status verified 2025-10

CONDITIONS: Normal Controls; MCI

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Normal Controls and MCI: All subjects will receive 18F-AV-1451 PET scan.
  Interventions: Drug: the radiotracer 18F-AV-1451

INTERVENTIONS:
Drug: the radiotracer 18F-AV-1451 — Subjects will receive a single IV bolus injection target dose of approximately 370 MBq (10 mCi ± 20%) of 18F-AV-1451 At approximately 75 minutes post dose, scanning will begin. An approximately 30-minute acquisition (six 5 minute intervals) will be performed

SUMMARY:
The purpose of this study is to measure the amount of a protein in the brain known as tau using an imaging procedure called Positron Emission Tomography (PET/CT). 18F-AV-1451 is a specialized radioactive PET imaging agent that is able to detect the presence of tau in the brain. In this study, the investigator will use the 18F-AV-1451 to capture images of tau in the brain. Findings from this study will likely provide insight into the mechanisms and distinctions of age-related cognitive decline and that of very early Alzheimer's disease.

DETAILED DESCRIPTION:
The investigator will conduct a tau PET scan in cognitively normal older adults enrolled in the National Alzheimer's Coordinating Center (NACC) study at the University of Pennsylvania's Penn Memory Center/Alzheimer's Disease Core Center (PMC/ADC).

Study Duration: Study duration will generally be a one-day study visit, but all subjects will be followed annually as part of their participation in the NACC study.

Participants may be asked to obtain a longitudinal follow-up scan approximately 2-3 years after the baseline scan.

Study Center(s): Penn Memory Center/Alzheimer's Disease Core Center at Perelman Center for Advanced Medicine, UPHS.

Objectives: To collect Tau PET imaging in cognitively normal older adults adults and patients with Mild Cognitive Impairment (MCI), in the NACC study to determine relationship to clinical, cognitive, and other biomarker data. In particular, the investigator will examine relationship of tau PET to structural and functional measures of medial temporal lobe (MTL) subregions. Findings from this study will likely provide insight into the mechanisms and distinctions of age-related cognitive decline and that of preclinical Alzheimer's Disease.

Number of Subject: 200, approximately 150 cognitively normal older adults and 50 with mild cognitive impairment.

Diagnosis and Main Inclusion Criteria Eligible subjects will be NACC cohort participants who have received a consensus conference designation of "Cognitively Normal and patients with Mild Cognitive Impairment (MCI)". All participants must have had their annual NACC clinical and cognitive examination within 6 months of the tau PET imaging and an MRI scan (including high resolution imaging of medial temporal lobe regions) and amyloid PET within 12 months.

Study Design: This is a cross-sectional study using the radiotracer 18F-AV-1451 to determine the relationship of tau pathology to both cross-sectional and longitudinal clinical and biomarker data of NACC cohort participants who are Cognitively Normal and patient with mild cognitive impairment . All subjects will already be part of the longitudinal cohort study, known as the "NACC" cohort, of the PMC/ADC. For the current protocol, participants will provide informed consent before beginning any study procedures. After screening assessments, participants will undergo PET scan imaging with 18F-AV-1451 and again 2 to 3 years after the baseline scan.

Study Drug Administration: Subjects will receive a single IV bolus injection target dose of approximately 370 MBq (10 mCi ± 20%) of 18F-AV-1451 At approximately 75 minutes post dose, scanning will begin. An approximately 30-minute acquisition (six 5 minute intervals) will be performed.

Adverse events will be monitored continuously during the imaging session. Subjects who experience any adverse event during an imaging session will not be discharged until the event has resolved or stabilized.

Statistical Methodology This is a data gathering protocol to obtain molecular imaging data in a cohort of older adults without cognitive symptoms. However, specific analyses will include quantitative measures of 18F-AV-1451 within the medial temporal lobe (MTL) and its relationship to volume and thickness of MTL subregions measured with high-resolution MRI. Additional correlation and regression analyses will be performed to determine relationships between 18F-AV-1451 and cross-sectional and longitudinal measures acquired as part of each individuals participation in the NACC longitudinal cohort study, including, but not limited to, MRI imaging, neurocognitive testing, demographic information, genetic data, and clinical outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Males and females ≥ 60 years of age.
2. Part of the NACC longitudinal cohort (Protocol #: 068200) of the PMC/ADCC with consensus conference designation of cognitively normal or MCI.
3. NACC longitudinal visit must be completed or scheduled to be completed within 6 months of the 18F-AV-1451 TAU PET scan.
4. A brain MRI must be performed within 12 months prior to their study scan date and be deemed of adequate quality that the scan may be used for study analysis, including 3T and/or 7 Tesla high-resolution imaging of medial temporal lobe structures.
5. An amyloid PET scan completed or scheduled within 12 months of their study scan date
6. Women must be post-menopausal or surgically sterile

Exclusion Criteria:

1. Any medical or psychiatric conditions that, in the opinion of the investigator, would compromise the subject's safety or successful participation in the study.
2. Have evidence of structural abnormalities such as major stroke or mass on MRI that is likely to interfere with analysis of the PET scan
3. Inability to tolerate or contraindication to imaging procedures in the opinion of an investigator or treating physician
4. Have current clinically significant cardiovascular disease .Have a history of significant or ongoing alcohol abuse or substance abuse or dependence based on medical record review or self-reported

Min Age: 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 200 cognitively normal older adults or patients with MCI
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2017-11-22 (Actual); Primary Completion 2025-10-08 (Actual); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Examine uptake of 18F-AV-1451 in the medial temporal lobe (MTL) and its relationship with high-resolution structural and functional MRI measures of MTL subregions. | 2 years.
  Specific analyses will include quantitative measures of 18F-AV-1451 within the medial temporal lobe (MTL) and its relationship to volume and thickness of MTL subregions measured with high-resolution MRI.

SECONDARY OUTCOMES:
Determine relationship to clinical, cognitive, and other biomarker data | 2 years.
  Correlation and regression analyses will be performed to determine relationships between 18F-AV-1451 and cross-sectional and longitudinal measures acquired as part of each individuals participation in the NACC longitudinal cohort study, including, but not limited to, MRI imaging, neurocognitive testing, demographic information, genetic data, and clinical outcomes.

CONTACTS AND LOCATIONS:
Overall Officials: David Wolk, MD, Principal Investigator — University of Pennsylvania
Locations (1):
- UPenn, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No